CLINICAL TRIAL: NCT01184820
Title: An Open-label Phase 1 Trial to Evaluate the Pharmacokinetics and Safety Profile of BAY94-9027 Following Single and Multiple Dose Administration in Two Cohorts of Previously Treated Male Subjects With Severe Hemophilia A
Brief Title: Trial to Evaluate the Pharmacokinetics and Safety Profile of BAY94-9027 Following Single and Multiple Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13401
Record Dates: First submitted 2010-07-13; First posted 2010-08-19 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Hemophilia A
Keywords: Pharmacokinetics; Safety
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Biological: BAY94-9027 + Recombinant Factor VIII (Kogenate FS, BAY14-2222)
- Arm 2 (Experimental)
  Interventions: Biological: BAY94-9027 + Recombinant Factor VIII (Kogenate FS, BAY14-2222))

INTERVENTIONS:
Biological: BAY94-9027 + Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Single dose of Kogenate FS and 16 doses of BAY94-9027 given 2 times a week for 8 weeks. Both drugs to be given intravenously.
  Arms: Arm 1
Biological: BAY94-9027 + Recombinant Factor VIII (Kogenate FS, BAY14-2222)) — Single dose of Kogenate FS and 9 doses of BAY94-9027 given once a week for 8 weeks. Both drugs to be given intravenously.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to describe the pharmacokinetics (PK) of BAY94-9027(the test drug). Pharmacokinetics means that we will measure how well the study drug corrects the factor VIII levels in your blood and how long it takes for the levels to fall back to your baseline level. The study is also designed to determine if the pharmacokinetics of BAY94-9027 change following repeat dosing over 8 weeks, determine if BAY94-9027 is safe, tolerable, and effective for the treatment of severe hemophilia A and define the appropriate dose of BAY94-9027. Two doses of BAY94-9027 will be studied.

The first 8 subjects enrolled in the study (cohort 1) will receive a low dose (25 IU/kg) and will be treated 2 days a week for 8 weeks (total of 16 doses). The second 8 subjects (cohort 2) will receive a higher dose and will be treated 1 day a week for 8 weeks (total 8 doses). All subjects will receive a single dose of rFVIII (Bayer Kogenate FS) to determine the PK by measuring blood levels for 2 days before they start the study drug BAY94-9027. Factor VIII blood levels for BAY94-9027 will be measured for 7 days after the first and last dose to see describe the PK. Safety & tolerability assessment include vital signs, coagulation and hematological parameter, clinical chemistry, measurement of FVIII inhibitor and polyethylene glycol (PEG) antibodies will be done during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with severe hemophilia A (documented plasma baseline Factor VIII level <1 %)
* >/= 18 but </= 65 years of age
* Previously treated with Factor VIII concentrate(s) for a minimum of 150 exposure days (as supported by the subject's medical history)
* Immunocompetent with a CD4+ lymphocyte count > 400/mm³
* Signed informed consent from subject

Exclusion Criteria:

* Documented history of inhibitor to Factor VIII with a titer >/= 0.6 BU (Biological Unit), by the Nijmegen modified assay. However, subjects with a maximum historical titer of </= 1.0 BU with the classical Bethesda assay on a single measurement but with at least 3 subsequent successive negative results (< 0.6 BU) thereafter are eligible.
* Unable to stop Factor VIII treatment to complete a minimum 72 hour washout
* Current evidence of inhibitor to Factor VIII with a titer >/= 0.6 BU, measured at the time of screening
* Abnormal renal function (serum creatinine > 1.5 times the upper limit of the normal range)
* Total bilirubin > 1.5 times the upper limit of the normal range
* Active hepatic disease (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels > 2 times the upper limit of the normal range)
* Any concomitant coagulation disorder other than hemophilia A (including lupus anticoagulant)
* Platelet count < 100,000/mm³
* Within the last 3 months prior to study entry or during the study will be treated with an immunomodulating drug other than anti-retroviral chemotherapy (e.g., a interferon, steroids, rituximab, etc)
* Any subject who requires major surgery during study period. Minor procedures may be approved if discussed in advance with the medical expert.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10-13 (Actual); Primary Completion 2011-10-10 (Actual); Study Completion 2011-10-10 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by measuring immunogenicity | Up to 8 weeks
  Antibodies to FVIII, polyethylene glycol (PEG) and BAY94-9027
Adverse events collection | Up to 8 weeks
Area under the plasma concentration vs time curve from time 0 to the last data point (AUC0-tlast) | Up to 8 weeks
Area under the plasma concentration vs time curve from zero to infinity after single (first) dose (AUC0-inf) | Up to 8 weeks
Maximum drug concentration in plasma (Cmax) | Up to 8 weeks
Half-life associated with the terminal slope (t1/2) | Up to 8 weeks
Time to reach maximum drug concentration in plasma after single (first) dose (Tmax) | Up to 8 weeks
Mean residence time (MRT) | Up to 8 weeks
Total body clearance (CL) | Up to 8 weeks
  Total body clearance of drug from plasma (volume/time) or (volume/time/body weight) or ((volume/time)*(1.73/body surface area)) calculated after intravenous administration
Apparent volume of distribution at steady state (Vss) | Up to 8 weeks
  Based on the chromogenic, one-stage and PEG capture assays
Incremental recovery of FVIII | Up to 8 weeks
  Recovery was assessed using two different assays (chromogenic and one-stage assay)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (4):
  - Davis, California
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Syracuse, New York

REFERENCES:
- [Result] Coyle TE, Reding MT, Lin JC, Michaels LA, Shah A, Powell J. Phase I study of BAY 94-9027, a PEGylated B-domain-deleted recombinant factor VIII with an extended half-life, in subjects with hemophilia A. J Thromb Haemost. 2014 Apr;12(4):488-96. doi: 10.1111/jth.12506. PMID 24843882